CLINICAL TRIAL: NCT04881266
Title: Long-Term Functional, Quality-of-Life, Neuropsychological and Cognitive Outcomes in COVID-19 Critical Illness Survivors
Acronym: LUNGTERMcov
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-00209
Record Dates: First submitted 2021-03-03; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Covid19; ARDS; Critical Illness; Neurocognitive Dysfunction
MeSH Terms: conditions — COVID-19; Critical Illness; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post Critical Illness due to COVID-19
- Caregivers of Post critically ill COVID-19 patients

SUMMARY:
The corona virus disease 2019 (COVID-19), suddenly incepted in December 2019 in Wuhan, China, leading to one of the greatest health care emergencies of the last century. Acute exacerbation of the COVID-19 can develop to an ARDS in a significant proportion of hospitalized cases, leading to invasive mechanical ventilation requirement and in some cases even mandating use of extra-corporeal membrane oxygenation. Being a disease having affected up to 15'581'009 as of July 25th, with more than 635'173 deaths, the long-term repercussions are of foremost importance. Health care systems world-wide will be faced with the aftermath of COVID-19, and optimal understanding of the long-term progression of COVID-19 may aid in a better care of critically ill patients and enable specifically targeted rehabilitation programs to improve outcomes.

Primary objective of this study is to assess the repercussions of COVID-19 induced critical illness on long-term functional status, quality-of-life, neuropsychology and cognition

DETAILED DESCRIPTION:
Health-care systems are ever improving, organ-support is advancing towards un-thought of possibilities and critical care medicine is becoming a field of evidence. As a consequence critical illness is bridgeable in many cases and intensive care unit (ICU) and hospital outcomes account for excellent survival numbers. In contrast to intensivist believes for decades nevertheless, a patient's life is not restored to normality the moment ICU survival is achieved, the real crucible is but starting at that moment. Sequela after critical illness are manifold and impact the functional status, quality-of-life, neuropsychology as well as cognition of patients surviving, leading to higher incidences of co-morbidities and a shortened life-expectancy.

Specifically reflecting the complex interplay between acute respiratory distress syndrome and long-term outcomes, the last decade has seen a plethora of research elaborating on the long-term outcomes of patients having suffered acute respiratory distress syndrome. The serious functional limitations in patients post critical illness were mainly linked to muscle wasting and weakness, and only secondarily to lung function, neuropathies and other etiologies. Further, the impaired neuropsychological status, especially mediated by posttraumatic stress disorder, and cognitive status have a great impact on the reduced health status and quality-of-life. On the other hand nevertheless, pulmonary function was near normal after up-to 5 years of follow-up. Finally, the impact of acute respiratory distress syndrome (ARDS) and critical illness have on caregivers should not be forgotten, with high levels of depressive symptoms having been reported.

Similar sequela were also described during the severe acute respiratory syndrome (SARS) epidemic in 2003.

The corona virus disease 2019 (COVID-19), suddenly incepted in December 2019 in Wuhan, China, leading to one of the greatest health care emergencies of the last century. Acute exacerbation of the COVID-19 can develop to an ARDS in a significant proportion of hospitalized cases, leading to invasive mechanical ventilation requirement and in some cases even mandating use of extra-corporeal membrane oxygenation. The median length of stay and of mechanical ventilation support in COVID-19 have been shown to be elevated in comparison to other ARDS etiologies. Being a disease having affected up to 92 million people during the year 2020, with more than 1.9 Million deaths reported, the long-term repercussions are of foremost importance. Health care systems world-wide will be faced with the aftermath of COVID-19, and optimal understanding of the long-term progression of COVID-19 may aid in a better care of critically ill patients and enable specifically targeted rehabilitation programs to improve outcomes.

The overall objective of this study is therefore to evaluate the long-term outcomes of COVID-19 induced critical illness regarding functional status, quality-of-life, neuropsychology and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Previous admission to one of the participating centers for COVID-19 critical illness treatment
* Previously proven SARS-CoV-2 infection
* Critical COVID-19 defined as respiratory failure and/ or shock and/ or multiorgan dysfunction or failure
* Signed Study Informed Consent

Exclusion Criteria:

* Age <18 years
* Rejection of the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The project population targeted with this research, consists of a post critically illness, COVID-19 diagnosed population having been admitted to one of the participating centers, as well as their closest caregiver. The closest caregiver is defined as the person spending most of the time with the patient and mainly responsible for the patients daily support and care (professional caregivers will not be included).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-07 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pulmonary Function: FEV1 | Mixed Model assessment of FEV1 over time at 3, 6 12 and 24 months post discharge from intensive care unit due to critical COVID-19
  Development of pulmonary function over time post intensive care unit stay due to COVID-19
Change in Quality of Life: SF-36 Score | Mixed Model assessment of SF-36 Score over time at 3, 6 12 and 24 months post discharge from intensive care unit due to critical COVID-19
  Development of quality of life over time post intensive care unit stay due to COVID-19
Change in Neuropsychological Status: RBANS Score | Mixed Model assessment of RBANS Score over time at 3, 6 12 and 24 months post discharge from intensive care unit due to critical COVID-19
  Development of Neuropsychological Status over time post intensive care unit stay due to COVID-19
Change in Quality of Life in Caregivers: SF-36 Score | Mixed Model assessment of SF-36 Score over time at 3, 6 12 and 24 months post discharge from intensive care unit due to critical COVID-19 of patients
  Development of quality of life in Caregivers over time post intensive care unit stay due to COVID-19 of patients

CONTACTS AND LOCATIONS:
Overall Officials: Reto A Schuepbach, Prof. Dr., Principal Investigator — Institute of Intensive Care Medicine, University Hospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided